CLINICAL TRIAL: NCT01531842
Title: Bacterial Resistance and Alterations in Conjunctival Flora Following Serial Intravitreal Injections
Brief Title: A Research Study to Evaluate the Effects of Repeated Intravitreal Injections on Bacteria Around the Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, Michele Formoso, Research Manager, Mid Atlantic Retina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#11-110
Record Dates: First submitted 2011-10-13; First posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Central Retinal Vein Occlusion; Choroidal Neovascularization; Age-related Macular Degeneration; Branch Retinal Vein Occlusion
Keywords: Conjunctival bacterial flora; prophylactic topical antibiotic; injection; intravitreal injection; bacterial resistance; serial injection; serial intravitreal injections; CNV; CRVO; AMD; BRVO
MeSH Terms: conditions — Retinal Vein Occlusion; Choroidal Neovascularization; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical antibiotic (Experimental): Patients will be randomized in a 1:1 fashion to receive a drop of topical antibiotic before and after the intravitreal injection in the +ABX arm (in addition to the typical prep with betadine).
  Interventions: Procedure: Conj flora Antibiotic resistance
- No Antibiotic Arm (Other): No topical antibiotics in the -ABX arm (only the typical prep with betadine)
  Interventions: Procedure: Conj flora Antibiotic resistance

INTERVENTIONS:
Procedure: Conj flora Antibiotic resistance — Patients will either receive a drop of topical antibiotic before and after the intravitral injection or no topical antibiotics (only typical prep with betadine).

SUMMARY:
This is a research study to evaluate the effects of repeated intravitreal injections on bacteria around the eye.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether conjunctival bacterial flora are altered and/or demonstrate increasing antibiotic resistance after serial intravitreal injections when a prophylactic topical antibiotic is used pre- and post-injection compared to when they are not used.

ELIGIBILITY:
Inclusion Criteria: Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Have been diagnosed with neovascular AMD, CRVO or BRVO.
* Have been determined by the investigator to require intravitreal injections of bevacizumab or ranibizumab.

Exclusion Criteria: Subjects meeting any of the following criteria are ineligible for study entry:

* Prior intraocular injection in either eye.
* Chronic use of opthalmic medication.
* Contact lens wear.
* Ocular surgery within the past 6 months.
* Use of ophthalmic medications in either eye or ocular infection within the past 6 months.
* Use of systemic antibiotics within 6 months.
* Known allergy or contraindication to povidone iodine or fluoroquinolones.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-02 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Determine if conj bacterial flora demonstrates increased antibiotic resistance if topical antibiotic used pre and post injection vs not used. | Prior to each of your eye injections for the first 4 injections and continue through the completion of your fourth injection, an anticipated maximum of 6 months.
  Evaluating the effects of repeated use of iodine drops with or without antibiotic eye drops on bacteria on the eye surface in patients undergoing injections in the eye to determine if conjunctival bacterial floar are altered or demonstate increasing antibiotic resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States